CLINICAL TRIAL: NCT05805514
Title: Improving Growth and Cognitive Development of the Disadvantaged Young Children by Providing Animal Source Food (ASF) and Psychosocial Stimulation in Resource Poor Setting
Brief Title: Improving Growth and Cognitive Development of the Disadvantaged Young Children in Resource Poor Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-22122
Record Dates: First submitted 2022-11-29; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: Complementary Feeding
Keywords: Child undernutrition; Cognitive development; Animal source food; Psychosocial stimulation; Complementary feeding; Nutrition education counselling

STUDY DESIGN:
Intervention Model Description: We will perform a post hoc test, which will enable us to examine the difference between various group means while simultaneously controlling for the family-wise error rate, to determine precisely which groups are distinct from one another. We will use linear mixed models for continuous outcomes (e.g. Bayley scores) and generalized linear mixed models for non-continuous outcomes (e.g. logistic mixed models for binary outcomes). Models will include a fixed effect, children as a random effect to account for the repeated measurements, and community-cluster as a random effect to account for the cluster effect. The models will be able to evaluate the impact of the interventions over time by testing for an interaction between time and intervention group. Analyses will be conducted to identify the baseline characteristics of mother-infant dyads who may benefit most from the intervention. Model assumptions will be checked and appropriate adjustments to the analysis will be made where necessary.
Who Masked: Outcomes Assessor
Masking Description: This is a community based randomized cobtrolled trial. Participants, care provider and investigator will know the intervention. Outcomes assessor (e.g. Anthrpometric measurer and psychosocial stimulation evaluator) will not know about the participant allocation and major outcome of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food and psychosocial intervention (Experimental): In Food and psychosocial intervention, the nutrition workers will be responsible for providing egg through food voucher, psychosocial stimulation, nutrition education counselling, child water, sanitation and hygiene message, and multiple micronutrient powder among the selected mothers/infant pairs.
  Interventions: Other: Animal source of food and psychosocial stimulation
- Food intervention (Experimental): In Food intervention, nutrition workers will give food egg, nutrition education counselling, water, sanitation and hygiene message, and multiple micronutrient powder among the selected mothers/infant pairs.
  Interventions: Other: Animal source of food
- Control (Placebo Comparator): In terms of control group, the nutrition workers will provide only nutrition education counselling among the selected mother-child pairs.
  Interventions: Other: Control

INTERVENTIONS:
Other: Animal source of food and psychosocial stimulation — 209 mother-child pair will receive the animal source of food and psychosocial stimulation for 12 months. Child will be recruited within 6-12 months.
  Arms: Food and psychosocial intervention
Other: Animal source of food — 209 mother-child pair will receive the animal source of food for 12 months. Child will be recruited within 6-12 months.
  Arms: Food intervention
Other: Control — 209 mother-child pair will receive the control package for 12 months. Child will be recruited within 6-12 months.
  Arms: Control

SUMMARY:
1. Burden:

   The period from birth to two years of age is the "critical window" for the promotion of optimal growth, health, and development. Insufficient quantities and inadequate quality of complementary foods, poor child-feeding practices and high rates of infections have a detrimental impact on growth. Approximately one-third of children less than five years of age in developing countries are stunted, and large proportions are also deficient in one or more micronutrients. An estimated six per cent or six hundred thousand under-five deaths can be prevented by ensuring optimal complementary feeding (CF) only.
2. Knowledge gap:

   The unprecedented global social and economic crisis triggered by the COVID-19 pandemic poses grave risks to the nutritional status and survival of young children in low-income and middle-income countries (LMICs) including Bangladesh. In this situation families living below the poverty line may unable to provide their children adequately for meeting their nutritional requirement. In the face of poverty, animal-sourced foods are the first to be dropped from children's diets though these are the most vital protein sources.
3. Hypothesis:

   An intervention package (child feeding counselling, food voucher for animal source food, WASH and micronutrient powder) will improve child growth (difference of 0.35 in mean Length-for-Age-Z-score) and cognitive outcome (difference of 3.80 in mean cognitive outcome) in the selected intervention area from rural Bangladesh compared to control area.
4. Objective:

   The general objective of this study is to evaluate an intervention package that should improve growth, cognitive development, appropriate complementary feeding practice, and water sanitation and hygiene (WASH) practices of children at risk of stunting in resource poor settings.
5. Methods:

We will use a community-based cluster randomized controlled three arms trial. The trial will be carried out in thirty clusters/wards (two to three villages making up each ward) within six unions of the Atpara Upazila in the Netrokona district. There will be three study groups (209 mothers/infant pairs in each treatment group I, II, and 209 mothers/infant pairs in the control group). The effect of the intervention package will be compared to the control group with similar population demography receiving only counselling on appropriate infant and young child feeding messages.

DETAILED DESCRIPTION:
Background:

Management of child malnutrition:

According to WHO report in 2003 Children over six months of age require up to 550 calories every day on top of being breastfed, traditional sources of which may cost up to BDT 40 (50 US cents. In Bangladesh, 2.87 million children under five are coming from the poorest segment (21.8% of the total population), this also includes 1.7 million children under five who belong to extremely poor households surviving on less than USD 1.9 per day (12.9% of the total population). For families surviving on less than USD 1.9 a day, the gross expenditure for their children's complimentary food would be one-fourth of their daily subsistence. This is surreal and unlikely to happen that these families will practice the recommended complementary feeding. As the cost of feeding one child is too high, these households are thus unable to provide their children adequately. In the face of poverty, animal-sourced foods are the first to be dropped from children's diets though these are the most crucial protein sources. There is a need to develop a strategy to support the cost of food supplement especially for children in this critical period what the proposed study is attempting.

Animal Source Food (ASF) Animal Source Foods are dense in a wide range of micronutrients linked to growth and cognitive development (iron, B12, choline), in addition to protein. World Health Organization (2014) described ASF as the best source of high-quality nutrient-dense food for 6-23 months of age children. One egg provides 57% of the RDA of protein and 98% of the adequate intakes (AI) of choline, 88% of vitamin B12, 25-50% of vitamin B6, folate and phosphorus, and 20% of zinc for 7-12-month-old children. Eggs also provide essential fatty acids, including DHA (22:6n-3), crucial for brain development, particularly during early life. This indicates the provision of eggs during the early complementary feeding period could promote cognitive development. Moreover, due to the COVID-19 pandemic, acute malnutrition among young children will be more pronounced due to an acute shortage of food and access to essential health and other services. It is assumed that stunting (chronic malnutrition) may fall back from the current level if no preventive measures have been taken.

Child Malnutrition and Cognitive Development:

Recently, the lancet series 2013 revealed that 165 million children with stunted growth had compromised cognitive development and physical capabilities and they were making yet another generation loss. In addition, undernutrition of children directly impacted a nation's economic advancement by at least 8% because of losses via poorer cognition and losses via reduced schooling. We have data showing a substantial deficit in development by 18 months of age and that stunting plays a significant role in producing this deficit in Bangladeshi children.

Nutrition counselling and ASF to improve growth and development of the children:

Study conducted by Ara et al, 2017 showed that nutrition education and counselling had a positive effect on initiation of breastfeeding within 1 hr of birth and exclusive breastfeeding practices thereafter for 6 months.

Sample size calculation:

The sample size based on LAZ is 135 and after considering 10% attrition, the total sample size is 202 per arm. We will however consider the largest sample size, which is 209. Since there will be three arms and a 1:1 ratio between the intervention and control, the overall sample size is 627.

Study sites:

The study will be conducted in one sub-district (Atpara) of the Netrokona district of Mymensingh division in Bangladesh. Population Total 132499 and main sources of income is Agriculture (76.46%). The prevalence of stunting and underweight in Netrokona is also high (>40% of children 12 - 24 months stunted).

Data collection tools:

Child growth: Trained research assistants will collect anthropometric measurements (weight and length) using established methods (Lohman 1992). The 2006 WHO Growth Standards will be used to construct anthropometric indices and standard WHO recommended indicators will be used to assess stunting (length-for-age <-2 Z score), wasting (weight-for-length <-2 Z score) and underweight (weight-for-age <-2 Z) where, z-score (observe value-mean value of reference population)/ SD value of reference population (WHO, 2006).

Child development: To measure home stimulation, family care indicators (FCIs) tools will be used to collect information on approaches that are employed by the family, such as toys, books, musical instruments at 6-23 months. Bayley Scales of Infant and Toddler Development-IV (38) will be used to assess child's critical developmental domains.

Home stimulation: The FCI contains five subscales: 'play activities' (PA), 'varieties of play materials' (VP), 'sources of play materials', 'household books', and 'magazines and newspapers' (MN). All subscales had acceptable short-term reliability. FCI will be assessed during baseline and end line.

Bayley Scales of Infant and Toddler Development™, Fourth Edition (Bayley™-4): Bayley Scales-4 will be used to assess child's three key developmental domains of cognition, language (expressive and receptive) and motor (fine and gross motor) at baseline and after 12 months. Bayley-4 used in previous studies in Bangladesh and has shown good inter-observer reliability and short-term test-re-test stability. Children's behavior using Wolke's Behaviour Rating Scale will also be measured at 12 months along with the Bayley test.

Child dietary diversity: Standard questions about infant feeding practices used in the Bangladesh DHS surveys (NIPORT 2017) will be used to monitor these patterns at the three-monthly data collection periods from enrolment till 12 months of intervention.

Child feeding practices: These will include questions about current breastfeeding status, current use of other liquids and solid foods, the timing of introducing different liquids or solid foods, use of bottles for feeding, and information about who is providing advice about infant feeding amongst family and friends. Trained interviewers will collect 24-hr dietary recalls using standard methods. All the foods consumed 24 hours prior to the interview will be recorded and portion sizes measured in local utensils. Recipes used to prepare foods will be recorded including the amounts of raw food used and the preparation methods.

Child mortality: A history of illnesses such as diarrhoea, dysentery (blood and/or mucus), fever and coughs, ear infections (purulent discharge) from the ears are obtained monthly using a 2-week recall method will be collected. These questions are based on the standard DHS infant morbidity recall questions expanded to include questions about ear discharge. Diarrhoea is defined as the passage of three or more loose or watery stools within the last 24 h. The presence of blood in the stools is defined as invasive diarrhoea. A single episode of diarrhoea lasting for more than two weeks is classified as persistent diarrhoea. Acute respiratory illnesses are defined as coughing with reported fast or rapid breathing or difficulty breathing, with or without fever.

Hand washing, food safety and structure observation: A questionnaire will be administered solely to assess core WASH indicators. Structured observations will be conducted quarterly to assess the regular hand-washing practices of mothers and children.

Household food security: The Household Food Insecurity Access Scale (HFIAS) and the Household Hunger Scale (HHS) will be used for measuring household food security (Coates et al., 2007). The HFIAS tool consists of nine questions to extract the information required for defining the household's food security status. Using those nine questions, household food insecurity status was categorized as food secure, mildly food insecure, moderately food insecure, or severely food insecure.

Intervention and evaluation plan:

There will be at least 20 visits by the nutrition workers (NWs). Team members from the icddr, b will organize and conduct hands-on training for all field staff who will be engaged with this project using the national Infant and Young Child feeding (IYCF) and basic training module and Reach Up early childhood parenting program.

1. ASF for food vouchers:

   Food voucher will be distributed to the mothers and caregivers to obtain ingredients for egg for children. Mothers will be advised to utilize the vouchers provided to purchase the egg. The field supervisor will provide each mother monthly food vouchers with an equivalent value of BDT 500/ month/child, exchanging for egg package from participating vendors without using cash. The research staff will monitor compliance. For programmatic reasons, the purchase will be restricted to specific food, and we will expect the voucher system will enable the program to have such control over the purchase.
2. Psychosocial stimulation (Early childhood developmental activities):

   Psychosocial stimulation intervention will include age-appropriate developmental messages, flip charts, and handmade toys provided by the NWs during home visits at regular intervals and feeding counseling. The mothers will be shown three to four age-appropriate stimulation activities with child and how to make toys using recycled materials. As children grow up, mothers will also be taught how to make simple one-page books, suitable for less literate mothers. The short version of the Stimulation Curriculum will take 30-40 minutes and will include the following activities during home visits:
   * Explaining 2-3 stimulation messages (e.g., how to show love, how to respond, how to facilitate communication etc.) along with their benefits on child development
   * Explaining 1 Pictorial Stimulation Calendar containing 3 to 4 age-appropriate activities with the child until next visit
   * Teaching mothers and other family members how to make toys from recycled materials
   * The performance of the NWs will be monitored at least four times during the study by the stimulation supervisors. Child developmental assessment will be done before and after 12 months of intervention.
3. Nutrition Education and Counselling (NEC):

   One NW will visit each participating mother-child pair at least two times per month to counsel the mothers to improve the children's dietary diversity. During counseling visits, particular emphasis will be given to feed the children the egg every day, provide appropriate amounts and frequencies of homemade complementary foods, and appropriate protein consumption from animal sources. NWs will use existing, harmonized BCC tools (NEC packages including flip charts, videos) to inform mothers about optimum child-feeding practices. The mothers will be encouraged to continue breastfeeding and support will be given for adequate frequency of complementary feeds and appropriate diversity foods. There will be further demonstrations of the preparation of complementary feeds as needed.
4. Multiple Micronutrient Powder (MNP):

   NWs will distribute a one-month supply of MNP (including iron, vitamin A, vitamin C, folic acid, zinc) during home visits to the mothers in the intervention area. They will instruct the mothers on mixing this micronutrient powder with the child's main meal by dividing the meal into two parts. Each child will be given fifteen sachets every month for a year. To ensure compliance, a re-sealable bag will be provided to every mother to store the empty powder sachets, which will be monitored monthly.
5. Maternal knowledge and practice: NWs will use existing and standardized questionnaire to collect data on infant and young child feeding practices, child care, early childhood development.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-15 months
2. Households having moderate to severe food insecurity
3. Households having monthly income < BDT 10,000
4. Households dependent on irregular income
5. Households have plan to stay in the study area for next 1 year
6. Households not involved with any nutrition or social safety net programme

Exclusion Criteria:

1. Children aged less than 6 months
2. Children aged more than 15 months
3. Households having regular income and monthly income is more than BDT 10000
4. Households involved in any nutrition or social safety net programme

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 627 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To change the nutritional status under-two (6-23 mo) year children (a difference of 0.35 SD in the length-for-age z-score) from food insecure, low-income families in rural Bangladesh after receiving comprehensive intervention for 12 months | Anthropometry will be collected in every three months till 12 months
  • Difference in length-for-age z-score after 12 months (length measured in centimeters) (intervention vs control)
To change the developmental outcome of the under-two (6-23 mo) year children | Child developmental assessment will be done before and after 12 months of intervention
  Differences in children's cognition, language (expressive and receptive), motor (fine and gross motor) and behavioural development will be assessed by Bayley Scales after 12 months (intervention vs control)

SECONDARY OUTCOMES:
To change the dietary diversity of the under-two (6-23 mo) year children | • Differences in percentage of children at 6, 9, 12 months who receive complementary feeds • Differences in percentage of children consuming foods from >4 food groups
  * Differences in percentage of children who receive solid, semi-solid or soft foods.
  * Differences in percentage of children consuming foods from >4 food groups
To change hand washing and sanitation practice | Hand washing and sanitation practice assessment will be done before and after 12 months of intervention
  • Difference in percentage of handwashing practice

CONTACTS AND LOCATIONS:
Overall Officials: Gulshan Ara, MSc, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Atpara, Netrakona, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Data records will be kept in locked file cabinets. However, records may be reviewed by representatives from the Research Review Committee and Ethical Review Committee of icddr, b.
  All study related documents will be kept in locked cabinets in locked rooms with limited access. Information in the electronic database established at icddr, b will be password-protected and access will be available only to authorized research team members. Any information printed from this database will be stored in locked files until its use is complete and then shredded.
  The study investigators are responsible for ensuring complete and accurate documentation for the study and for each subject, including medical records, records detailing each subject's progress through the study, laboratory reports, Case Report Forms (CRFs), signed informed consent forms, correspondence with IRB(s), adverse event reports, and information regarding subject discontinuation and completion of the study.

REFERENCES:
- [Result] World Health Organization, 2003. Complementary feeding: report of the global consultation, and summary of guiding principles for complementary feeding of the breastfed child.
- [Result] Ravi, S. and Engler, M., 2015. Workfare as an effective way to fight poverty: The case of India's NREGS. World Development, 67, pp.57-71.
- [Result] Walker, S., 2020. The Impact of Dietary Egg Intake on Metabolic Health in Food Insecure Households. University of Arkansas.
- [Result] Headey D, Hirvonen K, Hoddinott J. Animal Sourced Foods and Child Stunting. Am J Agric Econ. 2018 Jul 31;100(5):1302-1319. doi: 10.1093/ajae/aay053. PMID 33343003
- [Result] Innis SM. Dietary (n-3) fatty acids and brain development. J Nutr. 2007 Apr;137(4):855-9. doi: 10.1093/jn/137.4.855. PMID 17374644
- [Result] Horton, S. and Steckel, R.H., 2013. Malnutrition: global economic losses attributable to malnutrition 1900-2000 and projections to 2050. How Much Have Global Problems Cost the Earth? A Scorecard from 1900 to, 2050, pp.247-272.
- [Result] Hamadani JD, Tofail F, Hilaly A, Huda SN, Engle P, Grantham-McGregor SM. Use of family care indicators and their relationship with child development in Bangladesh. J Health Popul Nutr. 2010 Feb;28(1):23-33. doi: 10.3329/jhpn.v28i1.4520. PMID 20214083
- [Result] Wolke D, Skuse D, Mathisen B. Behavioral style in failure-to-thrive infants: a preliminary communication. J Pediatr Psychol. 1990 Apr;15(2):237-54. doi: 10.1093/jpepsy/15.2.237. PMID 2374078
- [Result] Ara G, Khanam M, Papri N, Nahar B, Kabir I, Sanin KI, Khan SS, Sarker MSA, Dibley MJ. Peer Counseling Promotes Appropriate Infant Feeding Practices and Improves Infant Growth and Development in an Urban Slum in Bangladesh: A Community-Based Cluster Randomized Controlled Trial. Curr Dev Nutr. 2019 Jun 18;3(7):nzz072. doi: 10.1093/cdn/nzz072. eCollection 2019 Jul. PMID 31334480
- [Result] Bayley, N., 2006. Bayley scales of infant and toddler development.